CLINICAL TRIAL: NCT03708289
Title: Prospective Evaluation of Body Composition, Bone Health and Hormonal Status After Initiation of an Integrase-inhibitor-based Anti-retroviral Therapy in Treatment-naïve HIV-1-infected Individuals
Brief Title: Body Composition, Bone Health and Hormonal Status in HIV-1-infected Individuals
Acronym: BONBO
Status: Terminated | Type: Observational
Why Stopped: recruitment slower than expected
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: UZB BONBO
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2016-09

CONDITIONS: HIV-1; Treatment-naïve
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: DXA scan — total and hip and spine dual energy x-ray absorptiometry
Other: Achilles bone US
Other: Medical body composition measurements
Other: Resting energy expenditure measurement

SUMMARY:
Improved survival of people living with HIV has resulted in an increased occurrence of other comorbidities, such as cardiovascular, renal, bone and endocrine pathologies.

The data that is currently available on cART-associated changes in bone mineral density, body composition and hormonal values is short-term and mainly derived from patients initiating cART in accordance with previous treatment guidelines. As current guidelines recommend earlier cART initiation and as PI-based regimens are becoming less frequently used, a favorable outcome on bone health, body composition measures and endocrine status might be expected.

This study will therefore prospectively document alterations in bone mineral density, body composition and endocrine status in HIV-infected patients in whom, in the current treatment era, an INSTI-based cART regimen is initiated as a first line regimen.

DETAILED DESCRIPTION:
Patients will be included at the initiation of cART. The follow up for this study is planned to fit within the routine follow up consultations and includes some extra experimental investigations, such as the medical body composition measurements, resting energy expenditure measurement, Achilles bone ultrasonometer and DXA scans. Standard blood and urine samples will be taken, including standard analyses and some extra analyses for the study.

Physical activity will be monitored for 5 consecutive days using a bracelet device while patients will be asked to record their food intake using a standardized diet agenda.

Total follow up time will be 144 weeks and includes 12 visits in total.

ELIGIBILITY:
Inclusion Criteria:

* Documented and confirmed HIV-1-infection
* Aged 18 years or above
* Naïve to anti-retroviral treatment, unless anti-retrovirals were taken in the context of occupational or non-occupational post-exposure prophylaxis or in the context of prevention of mother-to-child transmission
* Willingness to sign the written informed consent

Exclusion Criteria:

* Pregnancy and breastfeeding
* Patients receiving medical care through an 'emergency care package'

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected patients aged 18 years or more, antiretroviral treatment naïve
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in BMD from baseline | 144 weeks of follow-up
Assessment of changes in trunk fat from baseline | 144 weeks of follow-up
Determination of the incidence of subclinical and clinical hypothyroidism | Within 144 weeks of follow-up

SECONDARY OUTCOMES:
Correlation between T-scores obtained by Achilles bone ultrasonometer (screening tool) and hip and spine DXA scan (gold standard) | 144 weeks of follow-up
Correlations between changes in body composition and endocrine values | 144 weeks of follow-up
Correlation between changes in VAT and trunk fat and changes in waist circumference | 144 weeks of follow-up
Description of changes in body composition in relation to the resting energy expenditure | 144 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sabine D Allard, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No